CLINICAL TRIAL: NCT04652583
Title: Auricular Muscle Zone Stimulation for Parkinson Disease (Earstim-PD)
Brief Title: Auricular Muscle Zone Stimulation for Parkinson Disease
Acronym: Earstim-PD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stoparkinson Healthcare Systems LLC (Industry)
Collaborators: The Parkinson Study Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: STP-PD-004
Record Dates: First submitted 2020-11-10; First posted 2020-12-03 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Active Stimulation 20 minutes (Active Comparator): Intramuscular stimulation
  Interventions: Device: Earstim - Active Stimulation
- Active Stimulation 60 minutes (Active Comparator): Intramuscular stimulation
  Interventions: Device: Earstim - Active Stimulation
- Sham Stimulation 20 minutes (Sham Comparator): Muscle-free-zone stimulation
  Interventions: Device: Earstim - Sham Stimulation

INTERVENTIONS:
Device: Earstim - Active Stimulation — Intramuscular stimulation
  Arms: Active Stimulation 20 minutes; Active Stimulation 60 minutes
Device: Earstim - Sham Stimulation — Sham stimulation
  Arms: Sham Stimulation 20 minutes

SUMMARY:
A Multicenter, Randomized, Blinded, Electronic Device in Subjects with Parkison Disease.

DETAILED DESCRIPTION:
This study is a multi-center, prospective, randomized, double-blinded, sham-controlled, within-subject design, 3-treatment, 3-period cross-over study involving 38 subjects with Parkinson's Disease who have the wearing-off phenomenon on oral levodopa therapy. All participants will receive three treatments on different days, each with different stimulation conditions. All subjects will wear the Earstim device on the ear ipsilateral to the side of the body more affected by Parkinson's Disease for 120 minutes during each of the three treatment applications.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or female ≥18 years of age.
2. Subject has Parkinson's Disease and is on levodopa therapy.
3. Subject experiences OFF periods with an "ON" score ≥20% better than the OFF score as measured by the MDS-UPDRS motor score (MDS-UPDRS Part III).
4. The subject's daily "OFF" time duration is ≥2 hours per day.
5. The subject's Hoehn-Yahr stage when "OFF" must be less than Stage 4 (i.e., subject must be able to walk without the use of an assisted device, such as a cane or a walker).
6. Subject receives levodopa at least TID with a minimum of 100 mg levodopa administered with each dose.
7. Subject can tolerate 2 hours in an "OFF" period without requiring rescue medication.
8. Subject is willing and able to not change Parkinson's Disease medications or dosages during the up to 2 week study therapy period.
9. Subject is willing to provide Informed Consent to participate in the study.
10. Subject is willing and able to comply with all study procedures and required availability for study visits.

Exclusion Criteria:

1. Subject has a medical or psychiatric comorbidity that can compromise participation in the study.
2. Subject has cognitive dysfunction defined by a Montreal Cognitive Assessment (MoCA) score <24.
3. Subject has moderate levodopa-induced dyskinesias as indicated by a score >2 on items 4.1 and/or 4.2 in the MDS-UPDRS Part IV.
4. Subject has clinically significant depression as determined by the Beck Depression Inventory-II score >15.
5. Subject is pregnant as determined by a urine pregnancy test at the screening visit.
6. Subject is of childbearing potential and is not surgically sterilized or does not use a reliable measure of contraception.
7. Subject has a form of Parkinsonism other than Parkinson's Disease, such as Drug-induced Parkinsonism or Multiple System Atrophy.
8. Subject has an implanted deep brain stimulator (DBS).
9. Subject is receiving direct intestinal infusions of levodopa.
10. Subject has epilepsy.
11. Subject medications are anticipated to change during the two (2) week study period (Note: the study requires stable medications during the device testing period).
12. Subject has a cardiac pacemaker or defibrillator, bladder stimulator, spinal cord stimulator or other active electronic medical device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III (Motor Score) at 20 minutes | Baseline, 20 minutes after the stimulation is initiated
  The primary efficacy endpoint is the overall change from baseline to 20 minutes after onset of stimulation in MDS-UPDRS motor score (MDS-UPDRS Part III), comparing the sham arm vs the average 20-minute change of the 20-minute and 60-minute auricular stimulation. Each parkinsonian sign or symptom is rated on a 5-point Likert-type scale (ranging from 0 to 4), with higher scores indicating more severe impairment.

SECONDARY OUTCOMES:
Area Under Curve | 120 minutes after stimulation is initiated.
  The area under the curve (AUC) of change from prior to stimulation in MDS-UPDRS Part III total motor score over the entire 120 minute post-stimulation follow-up interval, comparing the sham treatment to the 20 and 60 minute treatments with auricular muscle zone stimulation by subject and by treatment group.
Maximal improvement in MDS-UPDRS motor score (MDS-UPDRS Part III) from prior to stimulation to any of the follow-up time points up to 120 minutes after onset of stimulation. | 120 minutes after stimulation is initiated.
  Maximal improvement in MDS-UPDRS motor score (MDS-UPDRS Part III) from prior to stimulation to any of the follow-up time points (20 ,40, 60, 90, and 120 minutes after onset of stimulation). Each parkinsonian sign or symptom is rated on a 5-point Likert-type scale (ranging from 0 to 4), with higher scores indicating more severe impairment
Patient Global Impression of Change (PGIC) scored by the subject prior to stimulation and at the follow-up time points up to 120 minutes after onset of stimulation. | 120 minutes after stimulation is initiated.
  Patient Global Impression of Change (PGIC) scored by the subject prior to stimulation and at the follow-up time points (20,40, 60, 90, and 120 minutes after onset of stimulation). Seven point Likert scale ranging from 1= much worse to 7= much better
Timed Get Up and Go test prior to stimulation and at the follow-up time points up to 120 minutes after onset of stimulation. | 120 minutes after stimulation is initiated.
  Timed Get Up and Go test prior to stimulation and at the follow-up time points (20 ,40, 60, 90, and 120 minutes after onset of stimulation).
Clinical Global Impression of Change (CGIC) prior to stimulation and at the follow-up time points up to 120 minutes after onset of stimulation. | Baseline, 120 minutes after stimulation is initiated.
  Clinical Global Impression of Change (CGIC) prior to stimulation and at the follow-up time points (20 ,40, 60, 90, and 120 minutes after onset of stimulation). Seven point Likert scale ranging from 1= much worse to 7= much better
Kinesia-ONE™ Variable: Finger Tapping Speed Score comparison between the three different treatments at the specified times of just before stimulation and at the follow-up time points up to 120 minutes after onset of stimulation. | 120 minutes after stimulation is initiated.
  Kinesia-ONE scores ranged from 0 to 4 (where 0 is normal and 4 represents severe abnormalities), with negative change from Baseline scores indicating improvement in disease symptoms.
Kinesia-ONE™ Variable: Rest Tremor Score comparison between the three different treatments at the specified times of just before stimulation and at the follow-up time points up to 120 minutes after onset of stimulation. | 120 minutes after stimulation is initiated.
  Kinesia-ONE scores ranged from 0 to 4 (where 0 is normal and 4 represents severe abnormalities), with negative change from Baseline scores indicating improvement in disease symptoms.
Kinesia-ONE™ Variable: Averaged Finger Tapping Speed and Resting Tremor Scores comparison between each study arm at the specified times of just before stimulation and at the follow-up time points up to 120 minutes after onset of stimulation. | 120 minutes after stimulation is initiated.
  The finger tapping speed scores and resting tremor scores were averaged and provided as one score ranging from 0 to 4 (where 0 is normal and 4 represents severe abnormalities), with negative change from Baseline scores indicating improvement in disease symptoms.
Kinesia-ONE™ Variable: Postural Tremor Score comparison between the three different treatments at the specified times of just before stimulation and at the follow-up time points up to 120 minutes after onset of stimulation. | 120 minutes after stimulation is initiated.
  Kinesia-ONE scores ranged from 0 to 4 (where 0 is normal and 4 represents severe abnormalities), with negative change from Baseline scores indicating improvement in disease symptoms.
Kinesia-ONE™ Variable: Finger Tapping Amplitude Score comparison between the three different treatments at the specified times of just before stimulation and at the follow-up time points up to 120 minutes after onset of stimulation. | 120 minutes after stimulation is initiated.
  Kinesia-ONE scores ranged from 0 to 4 (where 0 is normal and 4 represents severe abnormalities), with negative change from Baseline scores indicating improvement in disease symptoms.
Kinesia-ONE™ Variable: Hand Grasp Speed Score comparison between the three different treatments at the specified times of just before stimulation and at the follow-up time points up to 120 minutes after onset of stimulation. | 120 minutes after stimulation is initiated.
  Kinesia-ONE scores ranged from 0 to 4 (where 0 is normal and 4 represents severe abnormalities), with negative change from Baseline scores indicating improvement in disease symptoms.
Kinesia-ONE™ Variable: Hand Grasp Amplitude Score comparison between the three different treatments at the specified times of just before stimulation and at the follow-up time points up to 120 minutes after onset of stimulation. | 120 minutes after stimulation is initiated.
  Kinesia-ONE scores ranged from 0 to 4 (where 0 is normal and 4 represents severe abnormalities), with negative change from Baseline scores indicating improvement in disease symptoms.
Kinesia-ONE™ Variable: Rapid Alternating Movement Speed Score comparison between the three different treatments at the specified times of just before stimulation and at the follow-up time points up to 120 minutes after onset of stimulation. | 120 minutes after stimulation is initiated.
  Kinesia-ONE scores ranged from 0 to 4 (where 0 is normal and 4 represents severe abnormalities), with negative change from Baseline scores indicating improvement in disease symptoms.
Kinesia-ONE™ Variable: Rapid Alternating Amplitude Score comparison between the three different treatments at the specified times of just before stimulation and at the follow-up time points up to 120 minutes after onset of stimulation. | 120 minutes after stimulation is initiated.
  Kinesia-ONE scores ranged from 0 to 4 (where 0 is normal and 4 represents severe abnormalities), with negative change from Baseline scores indicating improvement in disease symptoms.
Kinesia-ONE™ Variable: Dyskinesia Score comparison between the three different treatments at the specified times of just before stimulation and at the follow-up time points up to 120 minutes after onset of stimulation. | 120 minutes after stimulation is initiated.
  Kinesia-ONE scores ranged from 0 to 4 (where 0 is normal and 4 represents severe abnormalities), with negative change from Baseline scores indicating improvement in disease symptoms.
Determination by the investigator of dyskinesia severity by MDS-UPDRS Part IV prior to stimulation and at the follow-up time points up to 120 minutes after onset of stimulation. | 120 minutes after stimulation is initiated
  Determination by the investigator of dyskinesia severity by MDS-UPDRS Part IV prior to stimulation and at the follow-up time points (20 ,40, 60, 90, and 120 minutes after onset of stimulation). dyskinesia severity is rated on a 5-point Likert-type scale (ranging from 0 to 4), with higher scores indicating more severe impairment
Determination by a consensus between subject and investigator of whether the subject is "OFF" or "ON" prior to stimulation and at the follow-up time points up to 120 minutes after onset of stimulation. | 120 minutes after stimulation is initiated.
  Determination by a consensus between subject and investigator of whether the subject is "OFF" or "ON" prior to stimulation and at the follow-up time points (20 ,40, 60, 90, and 120 minutes after onset of stimulation).
Change in mood as measured by the Depressed Mood Score from baseline to 120 minutes after onset of stimulation. | 120 minutes after stimulation is initiated.
  Change in mood as measured by the Depressed Mood Score in Part I of MDS-UPDRS from pre-stimulation to 120 minutes after onset of stimulation.
Change in mood as measured by the Anxiety Mood Score from baseline to 120 minutes after onset of stimulation. | 120 minutes after stimulation is initiated.
  Change in mood as measured by the Anxiety Mood Score in Part I of MDS-UPDRS from pre-stimulation to 120 minutes after onset of stimulation.
Change in subjects' sense of well-being as measured by an exploratory ordinal scale prior to stimulation and at the follow-up time points up to 120 minutes after onset of stimulation. | 120 minutes after stimulation is initiated.
  Change in subjects' sense of well-being as measured by an exploratory ordinal scale prior to stimulation and at the follow-up time points (20 ,40, 60, 90, and 120 minutes after onset of stimulation). Scores ranged from +3 to -3 (+3 represents more comfortable - much greater peace of mind; and -3 represents more uncomfortable and have a much greater worse peace of mind

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf O Cakmak, MD, PhD, Study Director — Stoparkinson Healthcare Systems LLC; Stanley Fahn, MD, Principal Investigator — H. Houston Merritt Professor of Neurology, Columbia University Medical Center
Locations (8):
- United States (8):
  - University of Southern California, Los Angeles, California
  - Rocky Mountain Movement Disorder's Center, PC, Englewood, Colorado
  - Parkinson Disease and Movement Disorder Center of Boca Raton, Boca Raton, Florida
  - University of Florida, Gainesville, Florida
  - Rush University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Kansas, Kansas City, Kansas
  - Booth Gardner Parkinson's Care Center, Kirkland, Washington

IPD SHARING:
Plan to Share IPD: No